CLINICAL TRIAL: NCT05790278
Title: Evaluating the Prevalence of Purpose-related Existential Distress Among 2 Clinical Populations Compared to a Normative Sample
Brief Title: Purpose in Life Survey
Acronym: PIL
Status: Enrolling by invitation | Type: Observational
Sponsor: Mary Radomski (Other)
Responsible Party: Sponsor-Investigator, Mary Radomski, Principal Investigator, Allina Health System
Organization: Allina Health System (Other)
Other Study IDs: 1920306
Record Dates: First submitted 2023-03-10; First posted 2023-03-30 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer; Traumatic Brain Injury
MeSH Terms: conditions — Breast Neoplasms; Brain Injuries, Traumatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adults with Early Stage Cancer
  Interventions: Other: Survey
- Adults with Traumatic Brain Injury
  Interventions: Other: Survey
- Health Control Adults
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Completion of a Purpose in Life Survey

SUMMARY:
At present, there is no empirical data that specifies the likely prevalence of purpose in life disruption among various clinical populations. Between one-third and one-half of cancer survivors report some degree of existential distress during or after their treatment, but these findings are not specific to the domain of purpose in life.

To address the aforementioned gap, we propose to conduct a survey study to determine the prevalence of purpose disruption in two clinical populations and determine if the prevalence of purpose disruption in these populations is different from that of a normative population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Stage 1, 2, 3 cancer
* Cancer types: breast cancer, non-Hodgkin's lymphoma; colorectal cancer
* Receiving oncology services or treatment through AHCI
* Have completed primary cancer treatment within the past 12 months
* Able to communicate in English;
* Able to see and read (with or without assistive devices);
* Has access to a device (computer, phone, tablet) and an email address;
* Access to an internet connection.
* Has a known email address (in EPIC) and/or home telephone number
* Adults who sustained a traumatic brain injury within the past 12 months.
* Attending the 2022 MN State Fair

Exclusion Criteria:

* Have declined consent for use of medical records in research during admission to AH facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who are either (1) healthy controls, (2) individuals with a qualifying cancer diagnosis, or (3) individuals with a qualifying Traumatic Brain Injury
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Purpose Status Question | Through Study Completion, about 15 minutes
  A single forced-choice self-report screener question that we developed in order to characterize existential distress related to purpose in life (PSQ: "Related to living with purpose in life, right now I am: moving backwards; stalled; figuring it out; moving forward on a path").

SECONDARY OUTCOMES:
Work and Adjustment Scale | Through Study Completion, about 15 minutes
  A 5-item self-report questionnaire to characterize functioning related to work, social life, leisure, home management, and relationships.
Meaning in Life Questionnaire | Through Study Completion, about 15 minutes
  A 10-item questionnaire designed to measure 2 dimensions of meaning in life: Presence of Meaning (how much respondents feel their lives have meaning) and Search for Meaning (how much respondents strive to find meaning and understanding in their lives).
Life Engagement Test | Through Study Completion, about 15 minutes
  A 6-item self-report questionnaire that captures the extent to which a person engages in activities that are personally valued.

CONTACTS AND LOCATIONS:
Overall Officials: Mary V Radomski, PhD, Principal Investigator — Allina Health - Courage Kenny Rehabilitation Institute
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No